CLINICAL TRIAL: NCT02884206
Title: A Multicenter, Randomized, Double-blind, Active-controlled Study to Evaluate the Effects of LCZ696 Compared to Valsartan on Cognitive Function in Patients With Chronic Heart Failure and Preserved Ejection Fraction
Brief Title: Efficacy and Safety of LCZ696 Compared to Valsartan on Cognitive Function in Patients With Chronic Heart Failure and Preserved Ejection Fraction
Acronym: PERSPECTIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696B2320; 2016-001254-17 (EudraCT Number)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: heart failure; cognition; positron emission tomography; magnetic resonance imaging; LCZ696; valsartan; Chronic heart failure; CHF
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 200 mg bid (Experimental): Patients who were able to tolerate the treatment during the single-blind treatment run-in epoch. Following the run-in period, patients randomized in this arm were given LCZ696 at 200 mg twice daily for three years
  Interventions: Drug: LCZ696; Drug: Placebo of Valsartan
- Valsartan 160 mg bid (Active Comparator): Patients who were able to tolerate the treatment during the single-blind treatment run-in epoch. Following the run-in period, patients randomized in this arm were given valsartan at 160 mg twice daily for three years.
  Interventions: Drug: Valsartan; Drug: Placebo of LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 50, 100, and 200 mg tablets taken orally twice daily with matching placebo for valsartan
  Arms: LCZ696 200 mg bid
Drug: Valsartan — Valsartan 40, 80, and 160 mg tablets taken orally twice daily with matching placebo for LCZ696
  Arms: Valsartan 160 mg bid
Drug: Placebo of LCZ696 — Placebo to match LCZ696 50 mg, 100 mg, and 200 mg tablets
  Arms: Valsartan 160 mg bid
Drug: Placebo of Valsartan — Placebo to match valsartan 40 mg, 80 mg, and 160 mg tablets
  Arms: LCZ696 200 mg bid

SUMMARY:
This study was a multi-center, randomized, double-blind, parallel group, active comparator trial designed to evaluate the overall effect of LCZ696 compared to valsartan on cognitive function as assessed by the CogState comprehensive cognitive battery in patients with Heart failure and preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
The Screening epoch of approximately 3 weeks was used to assess eligibility. Eligible patients then entered the single-blind treatment run-in epoch (Active Run-In Epoch), which was designed to assess patient's tolerability to study drug and to determine patients who were likely to stay on study drug for the duration of the trial. The treatment run-in consisted of valsartan 40 mg bid (if necessary), followed by valsartan 80 mg bid, and then followed by LCZ696 100 mg bid, over 3 to 8 weeks duration. Patients unable to tolerate either valsartan or LCZ696 at the prescribed doses during the treatment run-in were not eligible for randomization and were discontinued from the study.

At randomization (Visit 199/201), eligible patients were randomized 1:1 to receive either LCZ696 200 mg bid or valsartan 160 mg bid (double-blind period).

Patients who terminated the study early were expected, and were encouraged, to attend all the protocol specified study visits, to perform all measurements as stipulated in the visit schedule and to remain in follow up for the duration of the trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic heart failure with current symptoms NYHA class II-IV
* Left ventricular ejection fraction > 40%
* NT-proBNP >= 125 pg/mL at screening visit
* Patient with evidence of adequate functioning to complete study assessments

Key Exclusion Criteria:

* Patients with acute decompensated heart failure requiring augmented therapy with diuretics, vasodilators and/or inotropic drugs
* Acute coronary syndrome (including myocardial infarction (MI)), cardiac surgery, other major CV surgery, or urgent percutaneous coronary intervention (PCI), carotid surgery or carotid angioplasty, history of stroke or transient ischemic attack within the 3 months prior to Screening visit or an elective PCI within 30 days prior to Screening visit
* Patients with history of hereditary or idiopathic angioedema or angioedema related to previous ACEi or ARB therapies
* Patients who require treatment with 2 or more of the following: an ACEi, an ARB or a renin inhibitor
* Patients with one of the following:

  1. Patients with serum potassium >5.2 mmol/L (mEq/L) at Screening visit
  2. Patients with serum potassium >5.4 mmol/L (mEq/L) at any visit during run-in treatment period or at randomization visit
  3. Systolic blood pressure (SBP) ≥180 mmHg at Screening visit, or
  4. SBP <110 mmHg at Screening visit, or
  5. SBP <100 mmHg or symptomatic hypotension as determined by the investigator at Visit 103 or at randomization visit
  6. Body mass index (BMI) >45 kg/m^2
* Patients with

  1. known pericardial constriction, genetic hypertrophic cardiomyopathy, infiltrative cardiomyopathy
  2. hemodynamically significant obstructive valvular disease
* Life-threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and atrial fibrillation or flutter with a resting ventricular rate >110 beats per minute
* Inability to perform cognitive battery or other study evaluations based on significant motor (e.g. hemiplegia, muscular-skeletal injury) or sensory (blindness, decreased or uncorrected visual or auditory acuity) skill
* Clinically significant cerebral pathology for example large cerebral aneurysm or space occupying lesion that may impact cognition as assessed by central MRI reader
* Mini mental state examination score less than 24 at screening
* Patients with a clinical diagnosis of Alzheimer's disease or other dementia syndromes or any indication for or current treatment with cholinesterase inhibitors and/or another prescription AD treatment (e.g. memantine).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (124):
- United States (48):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Sun City West, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Danbury, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Edgewater, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Homestead, Florida
  - Novartis Investigative Site, Inverness, Florida
  - Novartis Investigative Site, Jacksonville Beach, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Eunice, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Kalispell, Montana
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Elmer, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oregon City, Oregon
  - Novartis Investigative Site, Springfield, Oregon
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Rock Hill, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Gonzales, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tacoma, Washington
- Argentina (5):
  - Novartis Investigative Site, Buenos Aires, ARG
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
- Australia (4):
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Milton, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Geelong, Victoria
- Novartis Investigative Site, Aalst, Belgium
- Bulgaria (2):
  - Novartis Investigative Site, Sofia, BGR
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
- Croatia (2):
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Zagreb
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Tourcoing
- Germany (14):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bitburg
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg
- Italy (8):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pisa, PI
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Netherlands (2):
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amsterdam
- Poland (7):
  - Novartis Investigative Site, Tarnów, Lesser Poland Voivodeship
  - Novartis Investigative Site, Krakow, Maloposkie
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
- South Korea (3):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Novartis Investigative Site, Basel, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Meselik, Eskişehir
  - Novartis Investigative Site, Sivas
- United Kingdom (9):
  - Novartis Investigative Site, Axbridge, Somerset
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 137 centers across 20 countries
Pre-assignment Details: A total of 1200 patients were screened. Of them, 706 patients entered the run-in period. Patients entered different parts of the treatment run-in phase based on their use of renin angiotensin system blockade medications at the time of enrolment (valsartan 40 mg bid (if necessary), followed by valsartan 80 mg bid, and then followed by LCZ696 100 mg bid, over 3 to 8 weeks duration)
Groups:
- Run-in Period: Treatment run-in consisted of valsartan 40 mg bid (if necessary), followed by valsartan 80 mg bid, and then followed by LCZ696 100 mg bid, over 3 to 8 weeks duration.
Period: Valsartan Run-in Period
Arm/Group | Run-in Period | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Started (Valsartan run-in) | 706 | 0 | 0
Completed | 659 | 0 | 0
Not Completed | 47 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Adverse Event | 31 | 0 | 0
Not completed — Patient/guardian decision | 9 | 0 | 0
Not completed — Protocol deviation | 4 | 0 | 0
Not completed — Non-compliance with study treatment | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: LCZ696 Run-in Period
Arm/Group | Run-in Period | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Started | 659 | 0 | 0
Completed | 592 | 0 | 0
Not Completed | 67 | 0 | 0
Not completed — Adverse Event | 38 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Patient/guardian decision | 16 | 0 | 0
Not completed — Protocol deviation | 6 | 0 | 0
Not completed — Non-compliance with study treatment | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Double-Blind Period
Arm/Group | Run-in Period | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Started | 0 | 295 | 297
Safety Set | 0 | 295 | 297
PET Substudy Set | 0 | 244 | 247
Completed | 0 | 251 | 237
Not Completed | 0 | 44 | 60
Not completed — Death | 0 | 28 | 39
Not completed — Patient/guardian decision | 0 | 10 | 13
Not completed — Lost to Follow-up | 0 | 4 | 4
Not completed — Physician Decision | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Non-compliance with study treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participants are based on the Randomized population, as primary and secondary analysis are based on the Randomized Set
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg Bid | Valsartan 160 mg Bid | Total
Number analyzed (Participants) | 295 | 297 | 592
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.27 (6.749) | 72.61 (7.043) | 72.44 (6.895)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 143 | 277
  Male | 161 | 154 | 315
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 273 | 271 | 544
  Asian | 11 | 12 | 23
  Black | 6 | 9 | 15
  Native American | 2 | 0 | 2
  Unknown | 1 | 2 | 3
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the CogState Global Cognitive Composite Score (GCCS)
Description: The CogState cognitive battery was composed of 7 tests, which were administered electronically by the patients at scheduled visits. For each test, a standardized z-score was calculated. The GCCS was the average of the non-missing individual test z-scores. A higher score indicated better cognitive function.
  CogState GCCS changes from baseline (randomization) were analyzed using a repeated measures ANCOVA in which treatment, age stratification factor, Mini mental state examination stratification factor, education level, Apolipoprotein E ε4 allele status, cerebrovascular disease burden at screening, visit and treatment-by-visit interaction are included as fixed-effect factor, and baseline (randomization) GCCS and visit-by- baseline GCCS as covariates with a common unstructured covariance matrix among visits between treatment groups. The analysis was based on a direct likelihood method with an assumption of Missing at random.
Time Frame: Baseline, month 36
Population: The overall number of participants analyzed represents the participants in the Safety Set (SAF) with non-missing value of CogState GCCS at both, baseline and month 36.
  The SAF comprised all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Global Cognitive Composite Score
Arm/Group | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Number analyzed (Participants) | 195 | 183
Global Cognitive Composite Score | -0.0902 (0.0372) | -0.0722 (0.0383)
Statistical Analysis 1: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Repeated measure ANCOVA; Test type: Non-Inferiority — To demonstrate non-inferiority that LCZ696 does not lead to a relevant decrease in cognition compared to valsartan at year 3, the lower bound of 95% CI does not include the pre-specified non-inferiority (NI) boundary (Cohen's D) of -0.3. An effect size of 0.3 in Cohen's D is generally considered as small; p = 0.7363, ANCOVA; LSM = -0.0180, 95% CI 2-sided [-0.1230 to 0.0870]; Cohen's D: -0.0277, 95% CI: -0.1101 to 0.0778

2. Secondary Outcome: Change From Baseline in Cortical Composite Standardized Uptake Value Ratio (SUVr)
Description: The effects of LCZ696 compared to valsartan on Aβ deposition in the brain over 3 years were evaluated in a subset of patients using amyloid positron emission tomography (PET) imaging by assessing the change from baseline in cortical composite SUVr. PET imaging was performed at selected PET-capable centers on all eligible patients participating in the substudy. Sites with patients performing the PET scan were a subset of the overall patient population and overall sites for the study.
  Change from baseline to 3 years was analyzed based on an ANCOVA model with treatment, age, MMSE, amyloid status (+ve/-ve) stratification factors, region, APOE4 status and cerebrovascular disease burden as fixed effects, with baseline SUVr and treatment-by-baseline SUVr interaction as covariates for each of these imputed datasets. Results were obtained by applying Rubin's rules on the estimates from the imputed datasets.
Time Frame: Baseline, month 36
Population: The overall number of participants analyzed represents the participants in the PET substudy set (PET) with non-missing value at both, baseline and month 36.
  The PET comprised SAF patients who participated in PET substudy and had non-missing baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: value ratio (SUVr)
Arm/Group | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Number analyzed (Participants) | 147 | 134
value ratio (SUVr)
  Global cortical composite | 0.0273 (0.0114) | 0.0564 (0.0101)
  Cingulum posterior composite | 0.0416 (0.0113) | 0.0876 (0.0109)
  Frontal lobe composite | 0.0218 (0.0117) | 0.0434 (0.0104)
  Parietal lobe composite | 0.0231 (0.0119) | 0.0532 (0.0104)
  Temporal lobe composite | 0.0249 (0.0110) | 0.0418 (0.0097)
  White matter composite | 0.0061 (0.0094) | -0.0072 (0.0083)
Statistical Analysis 1: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Multiple Imputation ANCOVA in Global cortical composite; Test type: Non-Inferiority — To show that the point estimate of SUVr difference in mean change over 3 years is in favor of LCZ696 and the non-inferiority is demonstrated, with the upper bound of the 95% CI excluding the NI boundary of 0.01; p = 0.0579, ANCOVA; Least Squares Mean = -0.0292, 95% CI 2-sided [-0.0593 to 0.0010]

3. Secondary Outcome: Change From Baseline in Individual Cognitive Domains
Description: The effects of LCZ696 compared to valsartan on the individual cognitive domains (memory, executive function, and attention) over 3 years were evaluated by assessing the individual components of the CogState cognitive battery. Composite scores for the 3 individual cognitive domains were generated by combining the standardized z-scores of selected tests from the CogState cognitive battery. Each composite score was the average of the non-missing individual test z-scores. A higher score indicated better cognitive function.
Time Frame: Baseline, month 36
Population: The overall number of participants analyzed represents the participants in the Safety Set (SAF) with non-missing value at both, baseline and month 36.
  The number analyzed per row represents the participants with a valid value for the corresponding domain.
Measure: Least Squares Mean (Standard Error); unit: Z-scores
Arm/Group | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Number analyzed (Participants) | 197 | 185
Z-scores
  Memory domain | -0.0573 (0.0477) | -0.0580 (0.0490)
  Executive function domain: number analyzed (Participants) | 196 | 184
  Executive function domain | -0.0375 (0.0480) | -0.0702 (0.0493)
  Attention domain: number analyzed (Participants) | 197 | 184
  Attention domain | -0.1836 (0.0614) | -0.0794 (0.0634)
Statistical Analysis 1: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Repeated measure ANCOVA for memory domain; Test type: Superiority; p = 0.9916, ANCOVA; Least Squares Mean = 0.0007, 95% CI 2-sided [-0.1339 to 0.1353]; Cohen's D: 0.0009; 95% CI: -0.0912 to 0.0922
Statistical Analysis 2: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Repeated measure ANCOVA for executive function domain; Test type: Superiority; p = 0.6348, ANCOVA; Least Squares Mean = 0.0327, 95% CI 2-sided [-0.1024 to 0.1677]; Cohen's D: 0.0391, 95% CI: -0.0727 to 0.1192
Statistical Analysis 3: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Repeated measure ANCOVA for attention domain; Test type: Superiority; p = 0.2403, ANCOVA; Least Squares Mean = -0.1042, 95% CI 2-sided [-0.2783 to 0.0700]; Cohen's D: -0.0967, 95% CI: -0.1542 to 0.0387

4. Secondary Outcome: Change From Baseline in the Summary Score of the Instrumental Activities of Daily Living (IADL)
Description: The effects of LCZ696 compared to valsartan on the changes in IADL over 3 years were evaluated by as assessing the Functional activities questionnaire (FAQ) summary scores.
  The FAQ is a 30-point questionnaire that is made up of 10 questions that reflect a patient's ability to perform activities of daily living and to function independently. A score of 0 represents no impairment and a score of 30 represents severe impairment.
Time Frame: Baseline, month 36
Population: The overall number of participants analyzed represents the participants in the Safety Set (SAF) with non-missing value at both, baseline and month 36.
Measure: Least Squares Mean (Standard Error); unit: FAQ scores
Arm/Group | LCZ696 200 mg Bid | Valsartan 160 mg Bid
Number analyzed (Participants) | 197 | 186
FAQ scores | 0.5983 (0.2064) | 0.7089 (0.2115)
Statistical Analysis 1: Comparison: LCZ696 200 mg Bid vs Valsartan 160 mg Bid; Repeated measure ANCOVA; Test type: Superiority; p = 0.7081, ANCOVA; Least Squares Mean = -0.1105, 95% CI 2-sided [-0.6906 to 0.4696]; Cohen's D: -0.0308, 95% CI: -0.1208 to 0.0820

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 37 months.
Description: The analysis considered patients in the Enrolled set (ENR) for AEs reported during the run-in epoch and Safety set (SAF) for reported AEs during the double-blind randomized treatment epoch.
Groups:
- Valsartan Run-in 40 mg Bid: Treatment run-in with valsartan 40 mg bid (if necessary)
- Valsartan Run-in 80 mg Bid: Treatment run-in with valsartan 80 mg bid
- LCZ696 Run-in 100 mg Bid: Treatment run-in with LCZ696 100 mg bid
Arm/Group | Valsartan Run-in 40 mg Bid | Valsartan Run-in 80 mg Bid | LCZ696 Run-in 100 mg Bid | LCZ696 200 mg Bid | Valsartan 160 mg Bid
All-Cause Mortality (participants affected / at risk) | 0/318 | 1/675 | 2/659 | 28/295 | 39/297
Serious Adverse Events (participants affected / at risk) | 3/318 | 6/675 | 27/659 | 145/295 | 161/297
Other Adverse Events (participants affected / at risk) | 40/318 | 76/675 | 136/659 | 238/295 | 245/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan Run-in 40 mg Bid (N=318) | Valsartan Run-in 80 mg Bid (N=675) | LCZ696 Run-in 100 mg Bid (N=659) | LCZ696 200 mg Bid (N=295) | Valsartan 160 mg Bid (N=297)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombasthenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 8 | 12
Acute right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2 | 3
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 3 | 5
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 14 | 11
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 1 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular dissociation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Cardiac amyloidosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 6
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 15 | 15
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 5 | 5
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 4 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 8 | 8
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 7 | 3
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3 | 7
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Chondrodermatitis nodularis chronica helicis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 2 | 2
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Epiretinal membrane (Eye disorders) | 0 | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2
Cardiac death (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 2 | 0
Death (General disorders) | 0 | 0 | 0 | 5 | 3
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 8 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2
Strangulated hernia (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 2 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 0 | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 4 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 3 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 2 | 3
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 4 | 4
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 10 | 9
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 5 | 5
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 6 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Auricular haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 7
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Angiocardiogram (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Catheterisation cardiac abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Rubulavirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 3
Viral test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 6
Benign hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Carcinoid tumour in the large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Endometrial stromal sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 1
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 4 | 3
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 3 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 3 | 6 | 5
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 6 | 6
Bladder mass (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2
Cystitis interstitial (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Central sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 9 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 2 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 5
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 3 | 5
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 3
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan Run-in 40 mg Bid (N=318) | Valsartan Run-in 80 mg Bid (N=675) | LCZ696 Run-in 100 mg Bid (N=659) | LCZ696 200 mg Bid (N=295) | Valsartan 160 mg Bid (N=297)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 24 | 21
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 6 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 16 | 12
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3 | 17 | 22
Bradycardia (Cardiac disorders) | 1 | 2 | 2 | 7 | 5
Cardiac failure (Cardiac disorders) | 1 | 0 | 2 | 14 | 25
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 3 | 10
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 18 | 6
Cataract (Eye disorders) | 0 | 1 | 1 | 6 | 8
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 12
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 13 | 19
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 6
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 6
Nausea (Gastrointestinal disorders) | 6 | 2 | 1 | 10 | 8
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 4 | 7
Asthenia (General disorders) | 0 | 2 | 3 | 7 | 13
Fatigue (General disorders) | 1 | 2 | 7 | 16 | 23
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 9 | 13
Oedema peripheral (General disorders) | 1 | 2 | 1 | 24 | 25
Pyrexia (General disorders) | 1 | 1 | 0 | 4 | 6
Bronchitis (Infections and infestations) | 0 | 4 | 3 | 18 | 13
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 12 | 5
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 8 | 9
Cystitis (Infections and infestations) | 0 | 0 | 1 | 6 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 6 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 6 | 6
Nasopharyngitis (Infections and infestations) | 0 | 5 | 8 | 26 | 25
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 8 | 11
Sinusitis (Infections and infestations) | 1 | 1 | 3 | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 13 | 6
Urinary tract infection (Infections and infestations) | 2 | 1 | 4 | 26 | 21
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 6 | 9
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 4 | 19 | 15
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 7 | 3
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 6 | 7
Blood creatinine increased (Investigations) | 0 | 2 | 4 | 9 | 7
Blood pressure increased (Investigations) | 0 | 1 | 2 | 4 | 12
Glomerular filtration rate decreased (Investigations) | 1 | 4 | 4 | 15 | 16
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 2 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 7 | 8
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 9 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 11 | 8 | 31 | 41
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 14 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 6 | 9
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 6
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 7 | 4
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 25 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 22 | 28
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 7 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 10 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 12 | 11
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 7
Dizziness (Nervous system disorders) | 5 | 4 | 11 | 28 | 31
Headache (Nervous system disorders) | 1 | 4 | 3 | 11 | 7
Syncope (Nervous system disorders) | 0 | 1 | 3 | 7 | 4
Depression (Psychiatric disorders) | 0 | 0 | 3 | 13 | 12
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 4 | 8
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 14 | 13
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 1 | 5 | 8
Haematuria (Renal and urinary disorders) | 0 | 2 | 1 | 10 | 8
Renal failure (Renal and urinary disorders) | 1 | 3 | 4 | 5 | 7
Renal impairment (Renal and urinary disorders) | 0 | 0 | 3 | 26 | 31
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 6 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 10 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 9 | 17 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 21 | 34
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3 | 9
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 6
Hypertension (Vascular disorders) | 0 | 2 | 2 | 21 | 31
Hypotension (Vascular disorders) | 9 | 10 | 24 | 68 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT02884206/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT02884206/SAP_001.pdf